CLINICAL TRIAL: NCT01077609
Title: Fluticasone Propionate Nasal Spray (Flixonase) Safety in Patients With Allergic Rhinitis Registered in the UK General Practice Research Database
Brief Title: Flixonase Safety in Patients With Allergic Rhinitis (AR)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111983; WE50002
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Intranasal steroids; beclometasone diproprionate; steroid-related outcomes
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Allergic rhinitis (AR) & Flixonase: Patients initiating treatment for allergic rhinitis on intranasal fluticasone propionate
  Interventions: Drug: Intermittent, sub-chronic and chronic Flixonase use
- AR & prescription for intranasal steroid other than Flixonase: Random sample of patients initiating treatment for allergic rhinitis with an intranasal steroid other than Flixonase
  Interventions: Drug: Intermittent, sub-chronic and chronic use of intranasal steroids other than Flixonase

INTERVENTIONS:
Drug: Intermittent, sub-chronic and chronic Flixonase use — Intermittent exposure episode is a series of fewer than four sequential prescriptions for Flixonase with gaps of no more than 60 days between any two. Sub-chronic use episode is a series of at least four and not more than eight sequential prescriptions for Flixonase with gaps of no more than 60 days between any two. Chronic use episode is a series of at least nine sequential prescriptions for Flixonase and gaps of no more than 60 days between any two. A span of at least 180 days must occur between the first and last prescription.
  Groups: Allergic rhinitis (AR) & Flixonase
Drug: Intermittent, sub-chronic and chronic use of intranasal steroids other than Flixonase — Intermittent exposure episode is a series of fewer than four sequential prescriptions for an intranasal steroid other than Flixonase with gaps of no more than 60 days between any two. Sub-chronic use episode is a series of at least four and not more than eight sequential prescriptions for an intranasal steroid other than Flixonase with gaps of no more than 60 days between any two. Chronic use episode is a series of at least nine sequential prescriptions for an intranasal steroid other than Flixonase and gaps of no more than 60 days between any two. A span of at least 180 days must occur between the first and last prescription.
  Groups: AR & prescription for intranasal steroid other than Flixonase

SUMMARY:
This is an inception cohort study that analyses data from an administrative medical records database. The two inception cohorts are: 1) patients initiated on intranasal FP and 2) patients initiated on another INS (not FP). The candidates for the inception cohorts did not use any intranasal steroid in the year prior to initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patient records dated between January 1990 - January 2002 were used to develop the overall study cohort. The cohort was composed of the following patients:

  1. All patients with at least one prescription for Flixonase
  2. A random sample of patients having at least one prescription for an INS other than Flixonase

Exclusion Criteria:

Patient-level exclusion

* Patients with less than 180 days of continuous eligibility before index date
* Patients who are under four years of age at index date
* Patients who are older than 85 years of age at index date

Episode-level exclusion

-When patient history was divided into Flixonase or other INS use episodes, patients with less than 120 days of eligibility after the last prescription in the episode Patients with an event of interest 180 days prior to patients' entry into the cohort or anytime prior to an episode index date were automatically excluded from the analysis of that event. This exclusion criterion was applied to rule out prevalent conditions.

Ages: 4 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The General Practice Research Database (GPRD). Patient records dated between January 1990 - January 2002 were used to develop the overall study cohort.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Steroid-related outcomes: Cataracts, Glaucoma, Nasal septum perforation, Hypercorticism, Adrenal insufficiency, Fractures (limited to hip, wrist and vertebral as proxies for osteoporosis), Otitis media, Sinusitis, Infectious complications of sinusitis | Exposure episodes are defined as any series of prescriptions filled within 60 days of one another. Observation periods capture incident events beginning with the first prescription in the episode and ending 120 days after the last fill date.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline